CLINICAL TRIAL: NCT07216118
Title: Optimizing Navigation for Wellness And Resources Utilization in Youth With Type 2 Diabetes
Brief Title: Pilot-Testing Strategies to Improve Outcomes for Youth With Type 2 Diabetes by Addressing Health-Related Social Needs
Acronym: ONWARD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Mary Ellen Vajravelu, MD, Assistant Professor, University of Pittsburgh
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY25030030; 1R01DK142766-01 (NIH)
Record Dates: First submitted 2025-10-09; First posted 2025-10-14 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-10

CONDITIONS: Diabetes in Adolescence; Type 2 Diabetes; Social Needs
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Community Health Workers

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Tailored Resources and Text Messages (Experimental): Tailored Resources AND Text Messages:
  Tailored Resources: Participants will be offered resource lists and warm referrals specific to health-related social needs (HRSN) on a screener. Their clinical team will be sent screener results and asked to talk about and address HRSN at the visit without additional guidance. Participants will be offered physical resources related to disclosed HRSN (e.g., food box for food insecurity).
  Text Messages: Participants will receive text messages once per month for 3 months. Messages will state that community-based resources to address HRSN are available if needed, with a link to opt-in to resource lists and warm referral links. Messages will include contact information for the study and clinical teams for optional HRSN discussion. Community Health Worker will not be assigned.
  Interventions: Behavioral: Tailored Resources; Behavioral: Text Messages
- Tailored Resources and Community Health Worker (Experimental): Tailored Resources AND Community Health Worker (CHW):
  Tailored Resources: Participants will be offered resource lists and warm referrals specific to health-related social needs (HRSN) on a screener. Their clinical team will be sent screener results and asked to talk about and address HRSN at the visit without additional guidance. Participants will be offered physical resources related to disclosed HRSN.
  CHW: Participants will be assigned a trained CHW to support connection with resources to address HRSN.
  Interventions: Behavioral: Tailored Resources; Behavioral: Community Health Workers (CHW)
- Universal Empowerment and Text Messages (Experimental): Assigned to Universal Empowerment AND Text Messages:
  Universal Empowerment: Regardless of disclosed health-related social needs (HRSN), participants will be offered physical resources and the opportunity to meet with a social worker. In place of screening results, the clinical team will be sent a message requesting that, when seeing the patient in clinic, they use the provided, easily accessible empowering script about HRSN.
  Text Messages: Participants randomized to text message will receive text messages once per month for 3 months. Messages will state that community-based resources to address HRSN are available if needed, with a link to opt-in to resource lists and warm referral links. Messages will include contact information for the study and clinical teams for optional HRSN discussion. Community Health Worker will not be assigned to participants.
  Interventions: Behavioral: Universal Empowerment; Behavioral: Text Messages
- Universal Empowerment and Community Health Worker (Experimental): Universal Empowerment AND Community Health Worker (CHW):
  Universal Empowerment: Regardless of disclosed health-related social needs (HRSN), participants will be offered physical resources and the opportunity to meet with a social worker. In place of screening results, the clinical team will be sent a message requesting that, when seeing the patient in clinic, they use the provided, easily accessible empowering script about HRSN.
  CHW: Participants will be assigned a trained CHW to support connection with resources to address HRSN.
  Interventions: Behavioral: Universal Empowerment; Behavioral: Community Health Workers (CHW)

INTERVENTIONS:
Behavioral: Tailored Resources — Participants will be offered resource lists and warm referrals specific to health-related social needs (HRSN) on a screener. Their clinical team will be sent screener results and asked to talk about and address HRSN at the visit without additional guidance. Participants will be offered physical resources related to disclosed HRSN (e.g., food box for food insecurity).
  Other Names: Tailored
  Arms: Tailored Resources and Community Health Worker; Tailored Resources and Text Messages
Behavioral: Universal Empowerment — Regardless of disclosed health-related social needs (HRSN), participants will be offered resource lists and warm referral links for food, housing, and transportation needs. At clinic visit, all will be offered physical resources and the opportunity to meet with a social worker. In place of screening results, the clinical team will be sent a message requesting that, when seeing the patient in clinic, they use the provided, easily accessible empowering script about HRSN.
  Other Names: Universal
  Arms: Universal Empowerment and Community Health Worker; Universal Empowerment and Text Messages
Behavioral: Text Messages — Participants will receive text messages once per month for 3 months. Messages will state that community-based resources to address health-related social needs (HRSN) are available if needed, with a link to opt-in to resource lists and warm referral links. Messages will include contact information for the study and clinical teams for optional HRSN discussion. Community Health Worker will not be assigned.
  Other Names: Text Only
  Arms: Tailored Resources and Text Messages; Universal Empowerment and Text Messages
Behavioral: Community Health Workers (CHW) — Participants will be assigned a trained CHW to support connection with resources to address HRSN.
  Other Names: CHW
  Arms: Tailored Resources and Community Health Worker; Universal Empowerment and Community Health Worker

SUMMARY:
The goal of this clinical trial is to pilot test different strategies to address health related social needs (HRSN) experienced by adolescent and young adult patients with type 2 diabetes and their families. The main questions it aims to answer are:

* How feasible are the strategies?
* How acceptable are the strategies?
* How reliably and consistently can the strategies be implemented?

Participants will:

Attend regularly scheduled diabetes clinic visits. Complete surveys and interviews. Be connected to community resources and organizations to help address HRSN.

ELIGIBILITY:
Adolescent-Caregiver Dyads will be recruited together.

Adolescent Inclusion Criteria:

* Age 13 to 22 years old
* known diagnosis of type 2 diabetes
* followed clinically at UPMC Children's Hospital of Pittsburgh
* able to provide assent/consent

Caregiver Inclusion Criteria:

* Adult (18 years or older) identifying as a primary caretaker of an adolescent or young adult with type 2 diabetes
* Has an adolescent/young adult who agrees to participate in the study
* able to provide consent

Exclusion Criteria:

* Inability to complete study questionnaires in English

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2028-04 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Acceptability of Intervention: Health-Related Social Needs Screener | 1-week after baseline
  4-item Acceptability of Intervention Measure; completed by all adolescents and caregivers. Questions are specific to acceptability of the screening questionnaire used to assess health-related social needs, with responses ranging from completely disagree to completely agree (5-point scale). A mean of 4 or higher indicates acceptability.
Feasibility of Intervention: Health-Related Social Needs Screener | 1-week after baseline
  4-item Feasibility of Intervention Measure; completed by all adolescents and caregivers. Questions are specific to feasibility of the screening questionnaire used to assess health-related social needs, with responses ranging from completely disagree to completely agree (5-point scale). A mean of 4 or higher indicates feasibility.
Acceptability of Intervention: Tailored Approach to Address Health-Related Social Needs | 1-week after baseline; 3 months; 6 months
  4-item Acceptability of Intervention Measure; completed by adolescents and caregivers assigned to arms using a tailored approach (not universal empowerment). Questions are specific to acceptability of the tailored approach used to address health-related social needs, with responses ranging from completely disagree to completely agree (5-point scale). A mean of 4 or higher indicates acceptability.
Feasibility of Intervention: Tailored Approach to Address Health-Related Social Needs | 1-week after baseline; 3 months; 6 months
  4-item Feasibility of Intervention Measure; completed by adolescents and caregivers assigned to arms using a tailored approach (not universal empowerment). Questions are specific to feasibility of the tailored approach used to address health-related social needs, with responses ranging from completely disagree to completely agree (5-point scale). A mean of 4 or higher indicates feasibility.
Acceptability of Intervention: Universal Empowerment Approach to Address Health-Related Social Needs | 1-week after baseline; 3 months; 6 months
  4-item Acceptability of Intervention Measure; completed by adolescents and caregivers assigned to arms using a universal empowerment approach (not tailored approach). Questions are specific to acceptability of the universal empowerment approach used to address health-related social needs, with responses ranging from completely disagree to completely agree (5-point scale). A mean of 4 or higher indicates acceptability.
Feasibility of Intervention: Universal Empowerment Approach to Address Health-Related Social Needs | 1-week after baseline; 3 months; 6 months
  4-item Feasibility of Intervention Measure; completed by adolescents and caregivers assigned to arms using a universal empowerment approach (not tailored approach). Questions are specific to feasibility of the universal empowerment approach used to address health-related social needs, with responses ranging from completely disagree to completely agree (5-point scale). A mean of 4 or higher indicates feasibility.
Acceptability of Intervention: Text Messages to Address Health-Related Social Needs | 1-week after baseline; 3 months; 6 months
  4-item Acceptability of Intervention Measure; completed by adolescents and caregivers assigned to arms using text messages without community health workers to support resource connection. Questions are specific to acceptability of the text messages without community health worker approach used to address health-related social needs, with responses ranging from completely disagree to completely agree (5-point scale). A mean of 4 or higher indicates acceptability.
Feasibility of Intervention: Text Messages to Address Health-Related Social Needs | 1-week after baseline; 3 months; 6 months
  4-item Feasibility of Intervention Measure; completed by adolescents and caregivers assigned to arms using text messages without community health workers to support resource connection. Questions are specific to feasibility of the text messages without community health worker approach used to address health-related social needs, with responses ranging from completely disagree to completely agree (5-point scale). A mean of 4 or higher indicates feasibility.
Acceptability of Intervention: Community Health Workers to Address Health-Related Social Needs | 1-week after baseline; 3 months; 6 months
  4-item Acceptability of Intervention Measure; completed by adolescents and caregivers assigned to arms using text messages with community health workers to support resource connection. Questions are specific to acceptability of community health workers in addition to text messages to address health-related social needs, with responses ranging from completely disagree to completely agree (5-point scale). A mean of 4 or higher indicates acceptability.
Feasibility of Intervention: Community Health Workers to Address Health-Related Social Needs | 1-week after baseline; 3 months; 6 months
  4-item Feasibility of Intervention Measure; completed by adolescents and caregivers assigned to arms using text messages with community health workers to support resource connection. Questions are specific to feasibility of community health workers in addition to text messages to address health-related social needs, with responses ranging from completely disagree to completely agree (5-point scale). A mean of 4 or higher indicates feasibility.
Fidelity of Intervention | 1-week after baseline; 3 months
  Investigator developed survey around receipt of intervention components including resources requested and used, community health worker interactions, and text message receipt; completed by adolescents and caregivers in all arms. Frequency and types of resources used, as well as community organizations with which respondents interacted will be reported. Frequency and duration of contact with community health workers will be reported for those assigned to arms using community health workers.

SECONDARY OUTCOMES:
Health-related social needs: Food Insecurity | Baseline, 3 months, 6 months
  5 items from the PhenX repository; completed by adolescents and caregivers. Food insecurity assessment includes 5 questions assessing presence and frequency of experiences consistent with food insecurity; responses include "often," "sometimes," or "never" as well as "yes" and "no." "Often," "sometimes," or "never" are scored as 1, 2, and 3 respectively, with yes=1 and no=2. The sum of affirmative responses ("often," "sometimes," "yes") is the raw score, with 0-1 indicating high or marginal food security, 2-4 low food security, 5-6 very low food security. Percentage of positive responses (food insecurity: marginal, low, or very low food security) will be reported.
Health-related social needs: Housing Insecurity | Baseline, 3 months, 6 months
  3 items from the PhenX repository; completed by adolescents and caregivers. Housing is assessed using 3 questions about living situation, stress related to rent/mortgage, and problems with housing; responses describing worry about losing a place to live or not having a steady place to live, as well as problems with housing, or always, usually, or sometimes worrying about not having enough money to pay rent or mortgage indicate positive housing insecurity. Percentage of positive responses (housing insecurity) will be reported.
Health-related social needs: Transportation Insecurity | Baseline, 3 months, 6 months
  4 items from the PhenX repository; completed by adolescents and caregivers. Transportation barriers assessment is 4 questions, with positive barriers indicated by responses of having "some" or "a lot" of trouble getting transportation to the clinic for visits or if respondents delay or miss appointments due to transportation problems. Percentage of positive responses (transportation insecurity) will be reported.
Connection with community health workers (CHW) | Baseline, 3 months, 6 months
  Investigator-developed survey around hours of connection with CHW, activities conducted with CHW, and resource connections made through CHW; completed by adolescents and caregivers assigned to CHW
Hemoglobin A1C | Baseline, 3 months, 6 months
  As measured during clinic visit; for adolescents only. Reported as %.
Body Mass Index | Baseline, 3 months, 6 months
  As measured at clinic visits; for adolescents only. Reported as kg/m2.
Diet quality | Baseline, 3 months, 6 months
  Automated self-administered 24-hour diet recall; Healthy Eating Index; completed by adolescents only. HEI is on a 100-point scale, with higher scores indicating higher diet quality.
Diabetes distress | Baseline, 3 months, 6 months
  Problem Areas in Diabetes Scale; completed by adolescents only. The 5-item scale includes a range of 5 responses, from "not a problem" (=0) to "serious problem" (=4). A total score of >=8 indicates possible diabetes related emotional distress.
Medication adherence | Baseline, 3 months, 6 months
  Investigator-developed survey of doses of diabetes medication missed; completed by adolescents only. Questions include the number of days that daily diabetes medications were taken in the past 7 days, as well as number of times in the past 4 weeks that weekly diabetes medications were taken. Respondents will be categorized into fully adherent if they report taking daily medications 6-7 days out of the past 7 days and weekly medications at least 3 out of 4 past weeks; for those taking both daily and weekly, both daily and weekly medication adherence criteria must be met for fully adherent classification. Those not "fully adherent" will be categorized as non-adherent.
Diabetes self-management | Baseline, 3 months, 6 months
  Treatment of Self-Regulation Questionnaire; adolescents only. This 15-item survey includes statements related to regular disease self-management and uses a 7-point scale ranging from "not true at all" (1) to "completely true" (7). Two subscales are included: Autonomous Regulation and Controlled Regulation. Scores are averaged for each subscale, with higher scores indicating higher level of endorsement of that regulatory style.
Social Support | Baseline, 3 months, 6 months
  Multidimensional Scale of Perceived Support Scale (Zimet, Dahlem, Zimet, Farley, 1988); completed by adolescents and caregivers. The 12-item survey includes a 7-item scale of response from "very strongly disagree" (1) to "very strongly agree" (7). There are 3 subscales to indicate significant other, family, and friends support. Responses will be averaged by subscale, with higher numbers indicating greater support. A total score (average of 12 response) will be reported.
Trustworthiness of Community Health Workers (CHW) | Baseline, 3 months, 6 months
  Adapted version of Trust in Physician Scale (adapted from Merenstein Z, Shuemaker JC, Phillips RL 2023) for CHW; completed by adolescents and caregivers assigned to CHW. This 11-item scale includes response options ranging from "strongly disagree" to "strongly agree", with items indicating mistrust reverse scored. Total and average scores will be reported, with higher scores indicating greater trust.
Trustworthiness of Healthcare System | Baseline, 3 months, 6 months
  Medical Mistrust Scale; completed by adolescents and caregivers. This 12-item scale includes 5 response options ranging from "strongly disagree" to "strongly agree". Higher scores indicate greater trustworthiness.

CONTACTS AND LOCATIONS:
Overall Officials: Mary Ellen Vajravelu, MD MSHP, Principal Investigator — University of Pittsburgh; Maya I Ragavan, MD MPH MS, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share de-identified individual-participant level (IPD) data including demographic and health-related social needs data from participant self-report, clinical laboratory and body mass index data upon reasonable request from investigators.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 3 years after the publication of results.
Access Criteria: Investigators must submit a proposal in writing that describes planned analyses, and a data sharing agreement with the University of Pittsburgh must be signed.